CLINICAL TRIAL: NCT06347185
Title: Simultaneous Care in Recurrent and/or Metastatic Head and Neck Cancer: the SupCare Study
Acronym: SupCare
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The necessary funding for this study was not secured
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EORTC-2236-HNCG-QLG
Record Dates: First submitted 2024-01-25; First posted 2024-04-04 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Head and Neck Neoplasms
Keywords: Quality of life
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Health Services Needs and Demand

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Active Comparator): The oncologist will be the main referral of the patient, deciding the therapeutic approach, the assessments requested, in terms of type of exams and timing and the need of possible further support from other expertise. The oncologist will base the choices also upon the results of the Liverpool Head and Neck Patient Concern Inventory (PCI-H&N) and the patient's preferences. At the end of the first oncological visit, the physician will be asked to predict the survival of the patient.
  Interventions: Procedure: Palliative care requested as needed, integrated with the standard oncologic care (reactive approach)
- Integrated Care (Experimental): Besides the oncology visit, patient will have the palliative care expert visit and follow up. The oncologist will define the therapeutic approach and the assessments requested, in terms of type of exams and timing. The palliative care clinician and the oncologist will judge the burden of symptoms and together they will propose the suggested interventions to relief the symptoms, with a particular attention to a validated instrument (the PCI-H&N) and patient priority questionnaire's results.
  Interventions: Procedure: Early palliative care, integrated with the standard oncologic care (proactive approach)

INTERVENTIONS:
Procedure: Early palliative care, integrated with the standard oncologic care (proactive approach) — Besides the Oncology visit, patient will have the palliative care expert visit and follow up (proactive approach). The oncologist will define the therapeutic approach and the assessments requested, in terms of type of exams and timing. The palliative care clinician and the oncologist will judge the burden of symptoms and together they will propose the suggested interventions to relief the symptoms, with a particular attention to the Liverpool Head and Neck Patient Concern Inventory (PCI-H&N) and patient priority questionnaire's results.
  Arms: Integrated Care
Procedure: Palliative care requested as needed, integrated with the standard oncologic care (reactive approach) — The oncologist will be the main referral of the patient, deciding the therapeutic approach, the assessments requested, in terms of type of exams and timing and the need of possible further support from other expertise (reactive approach). The oncologist will base the choices also upon the results of the PCI-H&N and the patient's preferences. At the end of the first oncological visit, the physician will be asked to predict the survival of the patient.
  Arms: Standard of Care

SUMMARY:
This is a late phase II, prospective, multicenter randomized study, to assess the value of early palliative care integrated with the standard oncologic care in patients with Recurrent Metastatic (RM) Head and Neck Cancer (HNC) proposed to first line palliative systemic treatment.

The study randomizes patients in a 1:1 fashion to standard oncologic care, in which the palliative care is requested as needed (reactive approach) or to early palliative care integrated with the standard oncologic care (proactive approach).

Standard of Care: the oncologist will be the main referral of the patient, deciding the therapeutic approach, the assessments requested, in terms of type of exams and timing and the need of possible further support from other expertise. The oncologist will base the choices also upon the results of the Liverpool Head and Neck Patient Concern Inventory (PCI-H&N) and the patient's preferences. At the end of the first oncological visit, the physician will be asked to predict the survival of the patient.

Integrated approach: Besides the Oncology visit, patient will have the palliative care expert visit and follow up. The oncologist will define the therapeutic approach and the assessments requested, in terms of type of exams and timing. The palliative care clinician and the oncologist will judge the burden of symptoms and together they will propose the suggested interventions to relief the symptoms, with a particular attention to a validated instrument (the PCI-H&N) and patient priority questionnaire's results.

Stratification Factors

* Institution
* Performance Status (PS) (0 vs 1-2)
* Presence of any caregiver at home
* Type of treatment (Immunotherapy alone vs any other combination)

Study duration: the total study duration is estimated at 36 months, with a total accrual time estimated to be 24 months from first patient in (FPI) and with an additional follow-up period of 12 months.

End of study occurs when all patients have completed their end of study visit and the study is mature for all analyses defined in the protocol and the database has been cleaned and frozen for these analyses.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* Histological diagnosis of HNC of epithelial origin. Any sub-site of head and neck is eligible except endocrine tumours such as thyroid and parathyroid cancer
* First diagnosis of recurrent disease and/or distant metastasis; with recurrent disease not amenable to salvage surgery or re-irradiation
* Patient candidate to any first line systemic treatment
* Life expectancy more than 3 months
* PS Eastern Cooperative Oncology Group (ECOG) ≤2
* Adequate cognitive and reading abilities.
* Availability of baseline scores for Emotional Functioning and Pain
* Patient agrees to complete questionnaires at week 6, 15, 24 and 52 after systemic treatment start
* Before patient 's enrolment, written informed consent must be given according to International Council for Harmonisation (ICH)/Good Clinical Practice (GCP), and national/local regulations.

Exclusion Criteria:

* Patients requiring a palliative care consultation right from the beginning of treatment
* Cutaneous primary cancer
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be assessed and discussed with the patient before the enrolment in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-09 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in emotional functioning and pain scores according to Item List (IL) 250 questionnaire at 15 weeks. | at 15 weeks
  To assess the added value of early palliative care integrated with the standard oncologic care as measured by the difference in mean change from baseline to 15 weeks between arms in patient reported emotional functioning and pain.
  Minimum = -100; Maximum = +100; higher means better outcome

SECONDARY OUTCOMES:
Change from baseline in emotional functioning and pain scores according to Item List 250 (IL250) questionnaire at 6 weeks, 24 weeks and 52 weeks. | at 6 weeks, 24 weeks and 52 weeks
  Evaluate the added value of early palliative care integrated with the standard oncologic care as measured by the difference in mean change from baseline at alternative timepoints between arms in patient reported emotional functioning and pain.
  Minimum = -100; Maximum = +100; higher means better outcome
Change from baseline in the selected Health Related Quality of Life (HRQoL) scales from the Item List 250 (IL250) questionnaire at 6 weeks, 15 weeks, 24 weeks and 52 weeks | at 6 weeks, 15 weeks, 24 weeks and 52 weeks
  Evaluate the change from baseline in supportive patient-reported symptom and functional outcomes at 6 weeks, 15 weeks, 24 weeks and 52 weeks.
  Minimum = -100; Maximum = +100; higher means better outcome
Number of unplanned visits to emergency room or specialist visits | up to 52 weeks
  Evaluate the frequency of the unplanned access to emergency room or specialist visits
Hospitalization due to treatment toxicities or tumour signs/symptoms, as evaluated by number of admissions and duration | up to 52 weeks
  Frequency of hospitalization due to adverse effects of treatment or due to tumour symptoms/signs
Identification of the rate of patients starting a new systemic treatment in the last three months of life | until 1 year from last patient enrolled
  Frequency of oncological treatments in last three months of life.
Rate of patients receiving systemic treatment in the last month of life | until 1 year from last patient enrolled
  Identification of the rate of patients receiving systemic treatment in the last month of life
Rate of patients with a tracheostomy performed in the last 3 months of life | until 1 year from last patient enrolled
  Identification of the rate of patients with tracheostomy performed in the last 3 months of life.
Rate of patients with gastrostomy performed in the last 3 months of life | until 1 year from last patient enrolled
  Identification of the rate of patients with gastrostomy performed in the last 3 months of life.
Caregiver/family members' satisfaction (FAMcare questionnaire) at 15 weeks | at 15 weeks
  Assessment of the caregiver/family members' satisfaction. Minimum = -99; Maximum = +99; higher means better outcome.
Overall Survival (OS) | until 1 year from last patient enrolled
  Overall Survival
Prediction error of survival (defined as the difference between actual survival (AS) of patients and clinician prediction of survival (CPS)) | until 1 year from last patient enrolled
  Accuracy of physician prediction of survival

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Bossi, MD, Principal Investigator — Istituto Clinico Humanitas; Kathy Taylor, MSc, Principal Investigator — Universitätsmedizin Mainz - Institut fuer Medizinische -Biometrie, Epidemiologie und informatik; Luigi Lorini, MD, Principal Investigator — Istituto Clinico Humanitas